CLINICAL TRIAL: NCT01877655
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 3 Trial to Evaluate the Protective Efficacy and Safety of a Therapeutic Vaccine, ASP0113, in Cytomegalovirus (CMV)-Seropositive Recipients Undergoing Allogeneic, Hematopoietic Cell Transplant (HCT)
Brief Title: A Study to Evaluate a Therapeutic Vaccine, ASP0113, in Cytomegalovirus (CMV)-Seropositive Recipients Undergoing Allogeneic, Hematopoietic Cell Transplant (HCT)
Acronym: HELIOS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 0113-CL-1004; 2013-000903-18 (EudraCT Number)
Record Dates: First submitted 2013-06-12; First posted 2013-06-14 (Estimated); Results first posted 2018-11-28 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Cytomegalovirus (CMV)-Positive Recipients; Allogeneic, Hematopoietic Cell Transplant (HCT)
Keywords: ASP0113; Cytomegalovirus (CMV); Hematopoietic Cell Transplant (HCT)

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ASP0113 (Experimental): Participants received 1 mL of 5 mg/mL of ASP0113 via intramuscular injection in the deltoid muscle alternating sides with each dose on days -14 to -3 pretransplant, 14 to 40, 60, 90 and 180 in relation to the day of transplant (Day 0).
  Interventions: Biological: ASP0113
- Placebo (Placebo Comparator): Participants received 1 mL of 5 mg/mL of matching placebo via intramuscular injection in the deltoid muscle alternating sides with each dose on days -14 to -3 pretransplant, 14 to 40, 60, 90 and 180 in relation to the day of transplant (Day 0).
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: ASP0113 — Intramuscular injection
  Arms: ASP0113
Drug: Placebo — Intramuscular injection
  Arms: Placebo

SUMMARY:
The purpose of the study was to evaluate the efficacy of ASP0113 compared with placebo as measured by a primary composite endpoint of overall mortality and CMV end organ disease (EOD) through 1 year post-transplant. Safety of ASP0113 in participants undergoing allogeneic HCT will also be evaluated.

DETAILED DESCRIPTION:
Participants will be followed for 5.5 years post-transplant for long-term safety via an annual telephone contact.

ELIGIBILITY:
Inclusion Criteria:

* Participant is a CMV-seropositive HCT recipient
* Participant is planned to undergo either of the following:

  * Sibling Donor Transplant
  * Unrelated Donor Transplant
* Participant has one of the following underlying diseases:

  * Acute myeloid leukemia (AML)
  * Acute lymphoblastic leukemia (ALL)
  * Acute undifferentiated leukemia (AUL)
  * Acute biphenotypic leukemia
  * Chronic myelogenous leukemia (CML)
  * Chronic lymphocytic leukemia (CLL).
  * A defined myelodysplastic syndrome(s) (MDS)
  * Primary or secondary myelofibrosis
  * Lymphoma (including Hodgkin's)

Exclusion Criteria:

* Participant has active CMV disease or infection or has received treatment for active CMV disease or infection within 3 months (90 days) prior to transplant
* Participant has a modified hematopoietic cell transplant comorbidity index (HCT-CI) score ≥ 4
* Participant has received a prior HCT and has residual Chronic Graft-versus-host Disease (cGVHD)
* Participant who is scheduled to have a cord blood transplant or a haploidentical transplant
* Participant has a platelet count of less than 50,000 mm3 within 3 days prior to randomization (platelet transfusions are allowed)
* Participant has aplastic anemia or multiple myeloma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 514 (Actual)
Dates: Start 2013-09-11 (Actual); Primary Completion 2017-09-28 (Actual); Study Completion 2022-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Global Development, Inc.
Locations (83):
- United States (27):
  - Site US10028, Birmingham, Alabama
  - Site US10044, Tucson, Arizona
  - Site US10035, San Francisco, California
  - Site US10026, Stanford, California
  - Site US10030, Tampa, Florida
  - Site US10012, Atlanta, Georgia
  - Site US10013, Chicago, Illinois
  - Site US10007, Indianapolis, Indiana
  - Site US10020, Westwood, Kansas
  - Site US10010, Louisville, Kentucky
  - Site US10043, Baltimore, Maryland
  - Site US10011, Baltimore, Maryland
  - Site US10021, Boston, Massachusetts
  - Site US10036, Rochester, Minnesota
  - Site US10042, St Louis, Missouri
  - Site US10023, Hackensack, New Jersey
  - Site US10047, New York, New York
  - Site US10027, Rochester, New York
  - Site US10025, Chapel Hill, North Carolina
  - Site US10016, Nashville, Tennessee
  - Site US10002, Dallas, Texas
  - Site US10045, Houston, Texas
  - Site US10046, Salt Lake City, Utah
  - Site US10031, Richmond, Virginia
  - Site US10039, Seattle, Washington
  - Site US10024, Seattle, Washington
  - Site US10019, Milwaukee, Wisconsin
- Australia (2):
  - Site AU43001, Herston, Queensland
  - Site AU43004, Adelaide, South Australia
- Belgium (3):
  - Site BE32001, Bruges
  - Site BE32005, Leuven
  - Site BE32007, Roeselare
- Canada (4):
  - Site CA15001, Vancouver, British Columbia
  - Site CA15002, Toronto, Ontario
  - Site CA15004, Montreal, Quebec
  - Site CA15003, Québec, Quebec
- France (4):
  - Site FR33011, Besançon
  - Site FR33005, Créteil
  - Site FR33009, Nantes
  - Site FR33010, Nice
- Germany (11):
  - Site DE49010, Bonn
  - Site DE49014, Cologne
  - Site DE49012, Düsseldorf
  - Site DE49013, Göttingen
  - Site DE49002, Leipzig
  - Site DE49015, Mainz
  - Site DE49007, Münster
  - Site DE49005, Stuttgart
  - Site DE49008, Tübingen
  - Site DE49006, Ulm
  - Site DE49001, Würzburg
- Japan (10):
  - Site JP81003, Nagoya, Aichi-ken
  - Site JP81011, Maebashi, Gunma
  - Site JP81007, Sapporo, Hokkaido
  - Site JP81010, Bunkyo-ku, Tokyo
  - Site JP81008, Chuo-ku, Tokyo
  - Site JP81009, Minato-ku, Tokyo
  - Site JP81004, Shinjuku-ku, Tokyo
  - Site JP81001, Fukuoka
  - Site JP81005, Fukuoka
  - Site JP81006, Osaka
- South Korea (4):
  - Site KR82004, Seoul, Seoul Teugbyeolsi
  - Site KR82002, Seoul
  - Site KR82003, Seoul
  - Site KR82001, Seoul
- Spain (10):
  - Site ES34001, Badalona
  - Site ES34006, Barcelona
  - Site ES34004, Barcelona
  - Site ES34005, Córdoba
  - Site ES34003, Granada
  - Site ES34011, Madrid
  - Site ES34007, Murcia
  - Site ES34010, Salamanca
  - Site ES34002, Santander
  - Site ES34009, Valencia
- Sweden (5):
  - Site SE46001, Gothenburg
  - Site SE46006, Linköping
  - Site SE46004, Lund
  - Site SE46003, Stockholm
  - Site SE46005, Umeå
- Taiwan (3):
  - Site TW88601, Taipei
  - Site TW88602, Taipei
  - Site TW88603, Taoyuan

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- [Derived] Ljungman P, Bermudez A, Logan AC, Kharfan-Dabaja MA, Chevallier P, Martino R, Wulf G, Selleslag D, Kakihana K, Langston A, Lee DG, Solano C, Okamoto S, Smith LR, Boeckh M, Wingard JR, Cywin B, Fredericks C, Lademacher C, Wang X, Young J, Maertens J. A randomised, placebo-controlled phase 3 study to evaluate the efficacy and safety of ASP0113, a DNA-based CMV vaccine, in seropositive allogeneic haematopoietic cell transplant recipients. EClinicalMedicine. 2021 Mar 19;33:100787. doi: 10.1016/j.eclinm.2021.100787. eCollection 2021 Mar. PMID 33842870
- See also: Link to results and other applicable study documents on the Astellas Clinical Trials website — https://www.clinicaltrials.astellas.com/study/0113-CL-1004/
- See also: Link to plain language summary of the study on the Trial Results Summaries website — https://ast.trialsummaries.com/Study/StudyDetails?id=14598&tenant=MT_AST_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 514 participants were enrolled across 11 countries. At least 30% of enrolled participants had cytomegalovirus (CMV) seronegative donor and underwent allogeneic hematopoietic cell transplant (HCT). After the primary study period (day 365) participants were monitored for 5.5 years post-transplant for long-term safety. After the primary period completion, 326 participants entered the long-term follow-up period.
Pre-assignment Details: Screening assessment occurred from 30 to 5 days before transplant. Participants who met the inclusion and none of the exclusion criteria were randomly assigned in a 1:1 ratio to receive either ASP0113 or placebo. The randomization to treatment was stratified by donor-recipient relatedness and by donor CMV serostatus.
Groups:
- ASP0113 5mg: Participants received 1 mL of 5 mg/mL of ASP0113 via intramuscular injection in the deltoid muscle alternating sides with each dose on days -14 to -3 pretransplant, 14 to 40, 60, 90 and 180 in relation to the day of transplant (Day 0).
Period: Overall Study
Arm/Group | Placebo | ASP0113 5mg
Started | 263 | 251
Received Treatment | 255 | 246
Completed | 165 | 154
Not Completed | 98 | 97
Not completed — Death | 57 | 52
Not completed — Withdrawal by Subject | 18 | 26
Not completed — Physician Decision | 11 | 10
Not completed — Miscellaneous | 4 | 4
Not completed — Randomized but Never Received Drug | 8 | 5

BASELINE CHARACTERISTICS:
Population: The analysis population was the All Randomized which consisted of all randomized participants whether they received study drug or not.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | ASP0113 | Total
Number analyzed (Participants) | 263 | 251 | 514
Age, Continuous [Mean (Standard Deviation); unit: Year] — Population: The analysis population was the all randomized.
  Year | 52.0 (13.15) | 51.8 (12.41) | 51.9 (12.78)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The analysis population was the all randomized.
  Participants
    Female | 105 | 110 | 215
    Male | 158 | 141 | 299
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: The analysis population was the all randomized.
  Participants
    Hispanic or Latino | 11 | 19 | 30
    Not Hispanic or Latino | 252 | 232 | 484
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: The analysis population was the all randomized.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 47 | 50 | 97
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 6 | 7 | 13
    White | 189 | 177 | 366
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 21 | 17 | 38
Strata [Count of Participants; unit: Participants] — Population: The analysis population was the all randomized.
  Participants
    Related Seropositive Donor | 65 | 73 | 138
    Related Seronegative Donor | 30 | 26 | 56
    Non-related Seropositive Donor | 96 | 73 | 169
    Non-related Seronegative Donor | 72 | 79 | 151
Primary Diagnosis [Count of Participants; unit: Participants] — Population: The analysis population was the all randomized.
  Participants
    Acute Myeloid Leukemia (AML) | 126 | 97 | 223
    Acute Lymphoblastic Leukemia (ALL) | 34 | 34 | 68
    Acute Undifferentiated Leukemia (AUL) | 1 | 2 | 3
    Acute Biphenotypic Leukemia (ABL) | 2 | 2 | 4
    Chronic Myelogenous Leukemia (CML) | 6 | 12 | 18
    Chronic Lymphocytic Leukemia (CLL) | 7 | 10 | 17
    Myelodysplastic Syndrome | 46 | 51 | 97
    Primary or Secondary Myelofibrosis | 8 | 11 | 19
    Lymphoma | 33 | 31 | 64
    Missing | 0 | 1 | 1
Conditioning Regimen [Count of Participants; unit: Participants] — Population: The analysis population was the all randomized.
  Participants
    Myeloablative | 122 | 120 | 242
    Non-Myeloablative | 131 | 124 | 255
    Missing | 10 | 7 | 17
Antithymocyte Globulin (ATG) Use [Count of Participants; unit: Participants] — Population: The analysis population was the all randomized.
  Participants
    Yes | 45 | 43 | 88
    No | 218 | 208 | 426
Height [Mean (Standard Deviation); unit: Centimeteres] — Population: The analysis population was the all randomized.
  Centimeteres | 170.6 (9.91) | 169.7 (9.88) | 170.2 (9.90)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Population: The analysis population was the all randomized.
  kg/m^2 | 27.0 (5.02) | 26.0 (5.05) | 26.5 (5.06)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Composite of All-Cause Mortality and Adjudicated Cytomegalovirus End Organ Disease (CMV EOD) Through 1 Year Post Transplant
Description: This was the composite of all-cause mortality and adjudicated CMV EOD through 1 year posttransplant, The CMV EOD was assessed by the independent and blinded adjudication committee, which counted events that were observed up to day 380 from transplantation. Deaths that occurred up to day 365 from transplant were also counted.
Time Frame: From first study dose injection (Day -14 to -3 prior to transplant) up to one year post study drug injection (Day 365)
Population: The analysis population was the full analysis set (FAS), which consisted of all randomized participants who received at least one dose of randomized study drug.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | ASP0113
Number analyzed (Participants) | 255 | 246
Percentage of Participants
  Participants With Composite Endpoint | 30.20 | 35.37
  All-Cause Mortality | 28.24 | 31.71
  Adjudicated CMV EOD | 3.53 | 6.10
Statistical Analysis 1: Comparison: Placebo vs ASP0113; Analysis of all-cause mortality and adjudicated CMV EOD. Analysis was completed using the Cochran-Mantel-Haenszel (CMH) test at the 1-sided 5% level stratified by use of antithymocyte globulin (ATG) and by receipt of a kidney from a living or deceased donor; Test type: Superiority; p = 0.205, Cochran-Mantel-Haenszel — P-value based on CMH general association test stratified by donor-recipient relatedness and donor CMV serostatus; Odds Ratio (OR) = 1.27, 95% CI 2-sided [0.87 to 1.85] — Odds ratio (ASP0113 vs placebo) and 95% CI was based on CMH general association test stratified by donor-recipient relatedness & donor CMV serostatus

2. Secondary Outcome: Percentage of Participants With Protocol-Defined CMV Viremia Through 1 Year Posttransplant
Description: Protocol-defined CMV viremia was defined as a CMV plasma viral load ≥1000 IU/mL as assessed by the central laboratory. Rate was based on cumulative incidence function estimated at 1 year. The central laboratory had the lower limit of quantification [LLOQ] for CMV viral load assessment, so when the viral load was below the LLOQ the actual viral load reading was not possible and was denoted as ≤LLOQ. If participant had any CMV viral load assessments greater than the LLOQ it was classified as viremic.
Time Frame: From first study dose injection (Day -14 to -3 prior to transplant) up to one year post study drug injection (Day 365)
Population: The analysis population was the FAS.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo | ASP0113
Number analyzed (Participants) | 255 | 246
Percentage of Participants | 58.6 [52.0 to 64.6] | 56.7 [50.1 to 62.8]
Statistical Analysis 1: Comparison: Placebo vs ASP0113; Analysis of CMV viremia through 1 year posttransplant. CMV viremia was defined by the protocol as CMV plasma viral load ≥ 1000 IU/mL as assessed by the central laboratory. The 95% CI was based on cumulative incidence function CMV viremia rate at 1 year; Test type: Superiority; p = 0.748, Cox Proportional Hazard Model — P-value based on cox proportional hazards model parameter estimate for the treatment effect; Parameter estimate from cox proportional hazard model (ASP0113 v placebo) with treatment & randomization strata adjusted for death as a competing risk; Hazard Ratio (HR) = 0.96, 95% CI 2-sided [0.76 to 1.22]

3. Secondary Outcome: Percentage of Participants With Adjudicated CMV-Specific Antiviral Therapy (AVT) Through 1 Year Posttransplant
Description: The CMV-specific AVT use was adjudicated by the independent and blinded committee. When the CMV-specific AVT was initiated, a central CMV viral load was obtained weekly until it was discontinued. Participants without any CMV-specific AVT events were censored on the last study evaluation.
Time Frame: From first study dose injection (Day -14 to -3 prior to transplant) up to one year post study drug injection (Day 365)
Population: The analysis population was the FAS.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo | ASP0113
Number analyzed (Participants) | 255 | 246
Percentage of Participants | 53.2 [46.8 to 59.1] | 54.6 [48.1 to 60.6]
Statistical Analysis 1: Comparison: Placebo vs ASP0113; Analysis of CMV-specific antiviral therapy (AVT) through 1 year. Time to first adjudicated CMV-specific therapy was defined as time to the start of AVT for CMV viremia. CMV-specific AVT was determined by the adjudication committee. Rate was based on cumulative incidence function estimate at 1 year; Test type: Superiority; p = 0.888, Cox Proportional Hazard Model — P-value based on cox proportional hazards model parameter estimate for the treatment effect; [statistical method as in outcome 2, analysis 1]; Hazard Ratio (HR) = 1.02, 95% CI 2-sided [0.80 to 1.29]

4. Secondary Outcome: Percentage of Participants With a Composite Endpoint of Protocol-defined CMV Viremia and Adjudicated CMV-Specific AVT Use
Description: Protocol-defined CMV viremia was as CMV plasma viral load ≥ 1000 IU/mL as assessed by the central laboratory. The CMV-specific AVT was determined by the adjudication committee. Participants with no posttransplant viral load data were excluded from the analysis.
Time Frame: From first study dose injection (Day -14 to -3 prior to transplant) up to one year post study drug injection (Day 365)
Population: The analysis population was the FAS.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | ASP0113
Number analyzed (Participants) | 255 | 246
Percentage of Participants | 60.78 | 60.98
Statistical Analysis 1: Comparison: Placebo vs ASP0113; Analysis of composite of CMV viremia and adjudicated CMV-AVT. The CMV viremia was defined by the protocol as CMV plasma viral load ≥ 1000 IU/mL as assessed by the central laboratory. CMV-specific AVT was determined by the adjudication committee. Participants with no posttransplant viral load data were excluded from the analysis; Test type: Superiority; p = 0.802, Cochran-Mantel-Haenszel — P value based on CMH general association test stratified by donor-recipient relatedness and donor CMV serostatus; Odds Ratio (OR) = 1.05, 95% CI 2-sided [0.73 to 1.51] — Odds ratio (ASP0113 vs placebo) and 95% CI based on CMH general association test stratified by donor recipient relatedness and donor CMV serostatus

5. Secondary Outcome: Percentage of Participants With First Occurrence of Adjudicated CMV-specific AVT or Adjudicated Diagnosis of CMV EOD After Study Drug First Injection Through 1 Year Posttransplant
Description: Rate was based on cumulative incidence function estimate at 1 year. Time to first CMV-specific AVT was defined as time to the start of AVT for CMV viremia or CMV EOD. CMV-specific AVT and EOD were determined by the adjudication committee. This endpoint was a composite endpoint based on the independent adjudication committee assessments of CMV-specific AVT and CMV EOD.
Time Frame: From first study dose injection (Day -14 to -3 prior to transplant) up to one year post study drug injection (Day 365)
Population: The analysis population was the FAS.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo | ASP0113
Number analyzed (Participants) | 255 | 246
Percentage of Participants | 54.4 [48.0 to 60.3] | 55.4 [48.9 to 61.5]
Statistical Analysis 1: Comparison: Placebo vs ASP0113; Analysis of rate of adjudicated CMV AVT or CMV EOD. Time to first CMV-specific AVT was defined as time to the start of AVT for CMV viremia or CMV EOD. CMV-specific AVT and EOD and were determined by the adjudication committee. Rate based on cumulative incidence function estimate at 1 year; Test type: Superiority; p = 0.928, Cox Proportional Hazards Model — P value based on cox proportional hazards model parameter estimate for the treatment effect; [statistical method as in outcome 2, analysis 1]; Hazard Ratio (HR) = 1.01, 95% CI 2-sided [0.80 to 1.28]

6. Secondary Outcome: All-Cause Mortality at 1 Year Posttransplant
Description: All-cause mortality through 1-year post-transplantation summary included all deaths and unknown survival status. For the known deaths, the adjudication committee assessed results and summarized them according to the following category: Mortality due to the participant's primary disease, and mortality due to causes unrelated to the participant's primary disease. Participants with unknown survival status at 1 year were considered dead for this analysis.
Time Frame: From first study dose injection (Day -14 to -3 prior to transplant) up to one year post study drug injection (Day 365)
Population: The analysis population was the FAS.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | ASP0113
Number analyzed (Participants) | 255 | 246
Percentage of Participants | 28.24 | 31.71
Statistical Analysis 1: Comparison: Placebo vs ASP0113; Analysis of all-cause mortality at 1 year. Participants with unknown survival status at 1 year were considered dead for this analysis; Test type: Superiority; p = 0.393, Cox Proportional Hazards Model — P value based on cox proportional hazards model parameter estimate for the treatment effect; Odds Ratio (OR) = 1.18, 95% CI 2-sided [0.81 to 1.73] — Odds ratio (ASP0113 vs placebo) and 95% CI based on CMH general association test stratified by donor-recipient relatedness and donor CMV serostatus

ADVERSE EVENTS:
Time Frame: All cause-Mortality: Baseline up to 5.5 years post transplant. Adverse Events: From first dose of study drug up to 30 days after last dose of study drug (Day 365).
Description: Treatment Emergent Adverse Event (TEAE) was defined as an adverse event observed after the first dose of study drug injection through Day 365 and within 30 days of the last dose of study drug. Drug-related TEAE was defined as any TEAE with at least possible relationship to study treatment as assessed by the investigator or with missing assessment of the causal relationship. AE data was not planned to be collected during the long-term follow-up period.
Arm/Group | Placebo | ASP0113 5mg
All-Cause Mortality (participants affected / at risk) | 100/255 | 105/246
Serious Adverse Events (participants affected / at risk) | 221/255 | 221/246
Other Adverse Events (participants affected / at risk) | 254/255 | 244/246
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=255) | ASP0113 5mg (N=246)
Agranulocytosis (Blood and lymphatic system disorders) | 3 (4) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 3 (4)
Aplasia pure red cell (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Bone marrow failure (Blood and lymphatic system disorders) | 1 (1) | 3 (3)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 11 (13) | 11 (14)
Haemolytic anaemia (Blood and lymphatic system disorders) | 2 (2) | 3 (3)
Haemolytic uraemic syndrome (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 5 (6) | 5 (6)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 3 (3)
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 3 (3) | 4 (5)
Cardiac failure (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac tamponade (Cardiac disorders) | 0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 2 (2) | 2 (2)
Pericarditis (Cardiac disorders) | 2 (2) | 1 (1)
Pulseless electrical activity (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Aural polyp (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Deafness neurosensory (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 (1) | 0 (0)
Mydriasis (Eye disorders) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 2 (3) | 2 (2)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anal fissure (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 11 (11) | 10 (13)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 2 (2)
Gastrointestinal toxicity (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Megacolon (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 8 (8) | 10 (10)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 2 (2) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 2 (2) | 1 (1)
Pneumatosis intestinalis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Proctalgia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 2 (2)
Small intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 7 (7) | 11 (12)
Asthenia (General disorders) | 2 (2) | 4 (4)
Chest pain (General disorders) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 3 (3)
Drug resistance (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 2 (2)
General physical health deterioration (General disorders) | 1 (1) | 0 (0)
Infusion site extravasation (General disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 1 (1) | 0 (0)
Mucosal inflammation (General disorders) | 2 (2) | 1 (1)
Multi-organ failure (General disorders) | 2 (2) | 6 (6)
Non-cardiac chest pain (General disorders) | 1 (1) | 1 (1)
Oedema due to cardiac disease (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 23 (29) | 26 (27)
Serositis (General disorders) | 0 (0) | 1 (1)
Sudden death (General disorders) | 1 (1) | 1 (1)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 2 (2)
Acute hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 2 (2) | 0 (0)
Hepatic vein occlusion (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 (2) | 2 (2)
Venoocclusive liver disease (Hepatobiliary disorders) | 4 (4) | 5 (5)
Acute graft versus host disease (Immune system disorders) | 9 (10) | 7 (7)
Acute graft versus host disease in intestine (Immune system disorders) | 76 (120) | 76 (123)
Acute graft versus host disease in liver (Immune system disorders) | 24 (30) | 18 (23)
Acute graft versus host disease in skin (Immune system disorders) | 122 (171) | 118 (165)
Alloimmunisation (Immune system disorders) | 1 (1) | 0 (0)
Chronic graft versus host disease (Immune system disorders) | 4 (5) | 2 (2)
Chronic graft versus host disease in intestine (Immune system disorders) | 6 (7) | 3 (3)
Chronic graft versus host disease in liver (Immune system disorders) | 7 (7) | 3 (3)
Chronic graft versus host disease in skin (Immune system disorders) | 5 (5) | 1 (1)
Abdominal abscess (Infections and infestations) | 1 (1) | 0 (0)
Abscess intestinal (Infections and infestations) | 1 (1) | 0 (0)
Acinetobacter bacteraemia (Infections and infestations) | 0 (0) | 2 (2)
Adenovirus infection (Infections and infestations) | 0 (0) | 1 (1)
Anorectal cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Aspergillosis (Infections and infestations) | 0 (0) | 1 (1)
Atypical mycobacterial infection (Infections and infestations) | 0 (0) | 1 (1)
Atypical pneumonia (Infections and infestations) | 1 (1) | 0 (0)
BK virus infection (Infections and infestations) | 2 (2) | 2 (2)
Bacteraemia (Infections and infestations) | 4 (4) | 4 (4)
Bacterial infection (Infections and infestations) | 0 (0) | 1 (1)
Bacterial sepsis (Infections and infestations) | 3 (4) | 3 (3)
Brain abscess (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 2 (2)
Bronchopneumonia (Infections and infestations) | 0 (0) | 1 (1)
Bronchopulmonary aspergillosis (Infections and infestations) | 3 (4) | 4 (4)
Campylobacter gastroenteritis (Infections and infestations) | 1 (1) | 1 (1)
Catheter site infection (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 3 (3)
Cerebral aspergillosis (Infections and infestations) | 1 (1) | 0 (0)
Citrobacter sepsis (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 5 (5) | 2 (2)
Clostridium difficile infection (Infections and infestations) | 4 (5) | 3 (3)
Corona virus infection (Infections and infestations) | 0 (0) | 2 (2)
Cystitis (Infections and infestations) | 1 (1) | 0 (0)
Cystitis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Cytomegalovirus colitis (Infections and infestations) | 1 (1) | 3 (3)
Cytomegalovirus gastritis (Infections and infestations) | 0 (0) | 2 (2)
Cytomegalovirus gastroenteritis (Infections and infestations) | 1 (1) | 1 (1)
Cytomegalovirus infection (Infections and infestations) | 6 (6) | 10 (10)
Cytomegalovirus viraemia (Infections and infestations) | 9 (11) | 11 (13)
Device related infection (Infections and infestations) | 2 (2) | 2 (2)
Device related sepsis (Infections and infestations) | 3 (3) | 0 (0)
Diarrhoea infectious (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Encephalitis cytomegalovirus (Infections and infestations) | 1 (1) | 0 (0)
Encephalitis herpes (Infections and infestations) | 0 (0) | 1 (1)
Encephalitis viral (Infections and infestations) | 0 (0) | 1 (1)
Enterococcal bacteraemia (Infections and infestations) | 2 (3) | 1 (1)
Enterococcal sepsis (Infections and infestations) | 2 (2) | 0 (0)
Enterocolitis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 2 (2)
Epstein-Barr viraemia (Infections and infestations) | 0 (0) | 1 (1)
Epstein-Barr virus infection (Infections and infestations) | 1 (1) | 1 (1)
Escherichia bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Escherichia sepsis (Infections and infestations) | 1 (1) | 3 (4)
Escherichia urinary tract infection (Infections and infestations) | 1 (1) | 2 (2)
Gangrene (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1)
Gastroenteritis adenovirus (Infections and infestations) | 1 (1) | 0 (0)
Genital herpes (Infections and infestations) | 0 (0) | 1 (1)
Hepatic candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Herpes simplex (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 5 (7) | 4 (4)
Herpes zoster ophthalmic (Infections and infestations) | 1 (1) | 1 (1)
Human herpesvirus 6 infection (Infections and infestations) | 2 (2) | 0 (0)
Human polyomavirus infection (Infections and infestations) | 0 (0) | 1 (1)
Infected skin ulcer (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 1 (1) | 2 (2)
Influenza (Infections and infestations) | 3 (3) | 3 (3)
Klebsiella bacteraemia (Infections and infestations) | 2 (2) | 1 (1)
Klebsiella sepsis (Infections and infestations) | 2 (2) | 2 (2)
Lobar pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Localised infection (Infections and infestations) | 1 (1) | 1 (1)
Lower respiratory tract infection bacterial (Infections and infestations) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 2 (3) | 4 (4)
Meningitis aseptic (Infections and infestations) | 0 (0) | 1 (1)
Neutropenic sepsis (Infections and infestations) | 1 (1) | 0 (0)
Oesophageal candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 2 (2) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1)
Peritonitis (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumocystis jiroveci pneumonia (Infections and infestations) | 2 (2) | 2 (3)
Pneumonia (Infections and infestations) | 15 (18) | 19 (20)
Pneumonia adenoviral (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia cytomegaloviral (Infections and infestations) | 1 (1) | 3 (3)
Pneumonia escherichia (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia fungal (Infections and infestations) | 2 (2) | 1 (1)
Pneumonia herpes viral (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia influenzal (Infections and infestations) | 2 (2) | 1 (1)
Pneumonia klebsiella (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia legionella (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia respiratory syncytial viral (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia staphylococcal (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia streptococcal (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia viral (Infections and infestations) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (2)
Pseudomonal bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Pulmonary mycosis (Infections and infestations) | 0 (0) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 2 (2) | 1 (1)
Respiratory tract infection (Infections and infestations) | 3 (3) | 4 (5)
Sepsis (Infections and infestations) | 20 (23) | 14 (14)
Septic shock (Infections and infestations) | 9 (10) | 10 (10)
Sialoadenitis (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 3 (3) | 1 (1)
Sinusitis fungal (Infections and infestations) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 4 (4) | 5 (6)
Staphylococcal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Streptococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Streptococcal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 0 (0)
Systemic mycosis (Infections and infestations) | 0 (0) | 1 (1)
Tubo-ovarian abscess (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 4 (4)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2)
Urinary tract infection bacterial (Infections and infestations) | 2 (2) | 3 (3)
Urinary tract infection enterococcal (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection fungal (Infections and infestations) | 0 (0) | 1 (1)
Viral haemorrhagic cystitis (Infections and infestations) | 2 (2) | 2 (2)
Viral infection (Infections and infestations) | 1 (1) | 0 (0)
Blood stem cell transplant failure (Injury, poisoning and procedural complications) | 4 (4) | 3 (3)
Drug dose omission (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (2)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Transfusion microchimerism (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Transplant failure (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1)
Computerised tomogram thorax abnormal (Investigations) | 1 (1) | 0 (0)
Immunosuppressant drug level increased (Investigations) | 1 (1) | 0 (0)
Liver function test abnormal (Investigations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 1 (3)
Transaminases increased (Investigations) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 1 (3)
Cachexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 4 (4) | 4 (4)
Diabetes mellitus (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myopathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Acute lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (3) | 0 (0)
Acute lymphocytic leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (8) | 5 (5)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 6 (6)
Acute myeloid leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 18 (21) | 17 (22)
Adult T-cell lymphoma/leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Central nervous system lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Chloroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Chronic lymphocytic leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (3)
Chronic myelomonocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Kaposi's sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (4)
Leukaemic infiltration brain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Monoclonal gammopathy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Mycosis fungoides recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 5 (5)
Myelofibrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Non-Hodgkin's lymphoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Peripheral T-cell lymphoma unspecified recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Post transplant lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2)
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
T-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
T-cell lymphoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
T-cell type acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Acute polyneuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Amnesia (Nervous system disorders) | 0 (0) | 1 (1)
Brain oedema (Nervous system disorders) | 0 (0) | 1 (1)
Central nervous system lesion (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Coma (Nervous system disorders) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 2 (2) | 3 (3)
Dizziness (Nervous system disorders) | 1 (1) | 2 (2)
Encephalitis (Nervous system disorders) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1) | 2 (2)
Facial paresis (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 2 (2)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Neurological decompensation (Nervous system disorders) | 1 (1) | 1 (1)
Paraplegia (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 2 (2)
Thalamus haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 2 (2)
VIIth nerve paralysis (Nervous system disorders) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 2 (2) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1) | 1 (1)
Disorientation (Psychiatric disorders) | 0 (0) | 1 (1)
Mania (Psychiatric disorders) | 0 (0) | 1 (1)
Mental disorder (Psychiatric disorders) | 1 (2) | 1 (1)
Mental status changes (Psychiatric disorders) | 2 (2) | 3 (3)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal colic (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 5 (6) | 3 (3)
Renal failure acute (Renal and urinary disorders) | 41 (46) | 28 (38)
Renal failure chronic (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal impairment (Renal and urinary disorders) | 2 (2) | 0 (0)
Renal injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal tubular necrosis (Renal and urinary disorders) | 1 (1) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (4)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Idiopathic pneumonia syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 3 (3)
Mediastinal mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Obliterative bronchiolitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 1 (1)
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 11 (13) | 8 (8)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Toxic epidermal necrolysis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (3)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Appendicectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Central venous catheter removal (Surgical and medical procedures) | 1 (1) | 0 (0)
Colectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Donor leukocyte infusion (Surgical and medical procedures) | 1 (1) | 0 (0)
Drug therapy (Surgical and medical procedures) | 0 (0) | 1 (1)
Stem cell transplant (Surgical and medical procedures) | 1 (1) | 2 (2)
Transurethral prostatectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 2 (2) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 3 (3) | 2 (2)
Microangiopathy (Vascular disorders) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1)
Thrombophlebitis (Vascular disorders) | 1 (1) | 0 (0)
Venoocclusive disease (Vascular disorders) | 1 (1) | 1 (1)
Venous thrombosis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=255) | ASP0113 5mg (N=246)
Anaemia (Blood and lymphatic system disorders) | 75 (160) | 66 (146)
Febrile neutropenia (Blood and lymphatic system disorders) | 92 (98) | 91 (101)
Leukopenia (Blood and lymphatic system disorders) | 23 (56) | 20 (51)
Neutropenia (Blood and lymphatic system disorders) | 65 (98) | 65 (99)
Pancytopenia (Blood and lymphatic system disorders) | 18 (19) | 21 (21)
Thrombocytopenia (Blood and lymphatic system disorders) | 48 (111) | 49 (131)
Tachycardia (Cardiac disorders) | 22 (24) | 22 (28)
Conjunctivitis (Eye disorders) | 17 (18) | 12 (12)
Dry eye (Eye disorders) | 37 (39) | 42 (45)
Abdominal discomfort (Gastrointestinal disorders) | 8 (11) | 13 (15)
Abdominal distension (Gastrointestinal disorders) | 22 (22) | 15 (18)
Abdominal pain (Gastrointestinal disorders) | 60 (83) | 62 (84)
Abdominal pain upper (Gastrointestinal disorders) | 33 (37) | 26 (32)
Constipation (Gastrointestinal disorders) | 103 (128) | 90 (119)
Diarrhoea (Gastrointestinal disorders) | 167 (244) | 166 (242)
Dry mouth (Gastrointestinal disorders) | 25 (31) | 30 (35)
Dyspepsia (Gastrointestinal disorders) | 25 (27) | 31 (35)
Gastritis (Gastrointestinal disorders) | 19 (19) | 19 (20)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 16 (17) | 24 (25)
Haemorrhoids (Gastrointestinal disorders) | 23 (26) | 27 (28)
Nausea (Gastrointestinal disorders) | 177 (261) | 178 (273)
Oral pain (Gastrointestinal disorders) | 16 (17) | 19 (20)
Proctalgia (Gastrointestinal disorders) | 20 (20) | 20 (23)
Stomatitis (Gastrointestinal disorders) | 69 (96) | 79 (105)
Vomiting (Gastrointestinal disorders) | 122 (178) | 125 (195)
Asthenia (General disorders) | 34 (43) | 30 (39)
Catheter site pain (General disorders) | 21 (23) | 22 (29)
Chills (General disorders) | 44 (59) | 36 (46)
Fatigue (General disorders) | 69 (80) | 58 (65)
Injection site erythema (General disorders) | 5 (5) | 49 (72)
Injection site induration (General disorders) | 3 (3) | 38 (57)
Injection site pain (General disorders) | 47 (83) | 193 (1053)
Injection site swelling (General disorders) | 4 (4) | 24 (36)
Malaise (General disorders) | 10 (11) | 15 (15)
Mucosal inflammation (General disorders) | 101 (147) | 75 (94)
Oedema (General disorders) | 21 (24) | 35 (39)
Oedema peripheral (General disorders) | 69 (95) | 66 (88)
Pain (General disorders) | 32 (34) | 27 (34)
Pyrexia (General disorders) | 128 (195) | 123 (180)
Hyperbilirubinaemia (Hepatobiliary disorders) | 16 (23) | 13 (17)
Chronic graft versus host disease (Immune system disorders) | 60 (109) | 62 (110)
Chronic graft versus host disease in intestine (Immune system disorders) | 21 (28) | 20 (22)
Chronic graft versus host disease in liver (Immune system disorders) | 35 (45) | 30 (43)
Chronic graft versus host disease in skin (Immune system disorders) | 46 (51) | 37 (40)
Engraftment syndrome (Immune system disorders) | 9 (9) | 13 (15)
Hypogammaglobulinaemia (Immune system disorders) | 19 (20) | 20 (20)
BK virus infection (Infections and infestations) | 13 (13) | 13 (15)
Clostridium difficile infection (Infections and infestations) | 16 (16) | 17 (18)
Cytomegalovirus infection (Infections and infestations) | 51 (64) | 45 (68)
Cytomegalovirus viraemia (Infections and infestations) | 96 (141) | 87 (132)
Device related infection (Infections and infestations) | 16 (16) | 16 (18)
Epstein-Barr virus infection (Infections and infestations) | 13 (15) | 15 (16)
Escherichia urinary tract infection (Infections and infestations) | 11 (11) | 13 (20)
Folliculitis (Infections and infestations) | 14 (18) | 8 (8)
Nasopharyngitis (Infections and infestations) | 12 (14) | 15 (15)
Oral candidiasis (Infections and infestations) | 27 (31) | 17 (18)
Oral herpes (Infections and infestations) | 17 (18) | 8 (13)
Pneumonia (Infections and infestations) | 13 (13) | 13 (13)
Staphylococcal bacteraemia (Infections and infestations) | 17 (20) | 20 (23)
Upper respiratory tract infection (Infections and infestations) | 27 (36) | 22 (24)
Fall (Injury, poisoning and procedural complications) | 10 (12) | 15 (17)
Alanine aminotransferase increased (Investigations) | 31 (47) | 33 (66)
Aspartate aminotransferase increased (Investigations) | 30 (45) | 30 (49)
Blood alkaline phosphatase increased (Investigations) | 17 (24) | 18 (23)
Blood bilirubin increased (Investigations) | 23 (48) | 21 (43)
Blood creatinine increased (Investigations) | 29 (42) | 22 (27)
Gamma-glutamyltransferase increased (Investigations) | 13 (24) | 15 (26)
Neutrophil count decreased (Investigations) | 33 (70) | 28 (62)
Platelet count decreased (Investigations) | 37 (83) | 28 (49)
Transaminases increased (Investigations) | 10 (11) | 18 (19)
Weight decreased (Investigations) | 15 (15) | 12 (15)
White blood cell count decreased (Investigations) | 23 (65) | 24 (45)
Decreased appetite (Metabolism and nutrition disorders) | 91 (109) | 72 (89)
Dehydration (Metabolism and nutrition disorders) | 13 (16) | 13 (31)
Diabetes mellitus (Metabolism and nutrition disorders) | 8 (8) | 17 (19)
Fluid overload (Metabolism and nutrition disorders) | 14 (14) | 11 (16)
Hyperglycaemia (Metabolism and nutrition disorders) | 66 (90) | 54 (81)
Hyperkalaemia (Metabolism and nutrition disorders) | 23 (40) | 30 (43)
Hyperuricaemia (Metabolism and nutrition disorders) | 10 (14) | 15 (17)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 30 (43) | 24 (53)
Hypocalcaemia (Metabolism and nutrition disorders) | 37 (58) | 28 (51)
Hypokalaemia (Metabolism and nutrition disorders) | 83 (120) | 92 (140)
Hypomagnesaemia (Metabolism and nutrition disorders) | 113 (157) | 113 (168)
Hyponatraemia (Metabolism and nutrition disorders) | 25 (42) | 26 (32)
Hypophosphataemia (Metabolism and nutrition disorders) | 27 (30) | 24 (28)
Arthralgia (Musculoskeletal and connective tissue disorders) | 27 (30) | 30 (42)
Back pain (Musculoskeletal and connective tissue disorders) | 39 (39) | 44 (52)
Bone pain (Musculoskeletal and connective tissue disorders) | 13 (14) | 10 (12)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 19 (25) | 14 (15)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 14 (15) | 10 (10)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 14 (14) | 19 (21)
Myalgia (Musculoskeletal and connective tissue disorders) | 19 (22) | 19 (23)
Neck pain (Musculoskeletal and connective tissue disorders) | 10 (10) | 16 (18)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 30 (31) | 32 (37)
Dizziness (Nervous system disorders) | 33 (38) | 33 (44)
Dysgeusia (Nervous system disorders) | 22 (22) | 23 (24)
Headache (Nervous system disorders) | 103 (153) | 103 (150)
Neuropathy peripheral (Nervous system disorders) | 17 (17) | 14 (17)
Tremor (Nervous system disorders) | 46 (49) | 23 (24)
Anxiety (Psychiatric disorders) | 44 (53) | 40 (42)
Depression (Psychiatric disorders) | 18 (18) | 11 (11)
Insomnia (Psychiatric disorders) | 76 (85) | 72 (86)
Dysuria (Renal and urinary disorders) | 29 (33) | 20 (25)
Haematuria (Renal and urinary disorders) | 15 (15) | 7 (8)
Pollakiuria (Renal and urinary disorders) | 14 (16) | 8 (9)
Renal failure (Renal and urinary disorders) | 16 (17) | 17 (19)
Cough (Respiratory, thoracic and mediastinal disorders) | 60 (71) | 55 (71)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 44 (53) | 40 (50)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 23 (28) | 34 (37)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 20 (21) | 22 (24)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 10 (12) | 17 (21)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 18 (20) | 8 (8)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 41 (42) | 30 (33)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 16 (17) | 18 (19)
Drug eruption (Skin and subcutaneous tissue disorders) | 30 (32) | 29 (31)
Dry skin (Skin and subcutaneous tissue disorders) | 20 (20) | 25 (26)
Erythema (Skin and subcutaneous tissue disorders) | 28 (37) | 34 (50)
Pruritus (Skin and subcutaneous tissue disorders) | 67 (85) | 59 (67)
Rash (Skin and subcutaneous tissue disorders) | 52 (61) | 51 (67)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 13 (17) | 12 (15)
Hypertension (Vascular disorders) | 83 (96) | 66 (78)
Hypotension (Vascular disorders) | 36 (37) | 39 (50)

LIMITATIONS AND CAVEATS:
In Oct 2014 data monitoring committee informed Astellas of the results of the first futility analysis. The FDA considered data for 68 participants included in futility analysis compromised and asked that it is not included in final efficacy analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data. Sponsor must receive a site's manuscript prior to publication for review and comment as specified in the Investigator Agreement.

DOCUMENTS (2):
  • Study Protocol (2016-10-28): https://cdn.clinicaltrials.gov/large-docs/55/NCT01877655/Prot_000.pdf
  • Statistical Analysis Plan (2017-05-19): https://cdn.clinicaltrials.gov/large-docs/55/NCT01877655/SAP_001.pdf